CLINICAL TRIAL: NCT05969548
Title: Personalized Brain Functional Sector-guided Continuous Theta Burst Stimulation Therapy at Different Doses for Aphasia After Stroke: a RCT
Brief Title: pBFS-guided cTBS at Different Doses for Aphasia After Stroke
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Changping Laboratory (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CPSA08HN60
Record Dates: First submitted 2023-07-23; First posted 2023-08-01 (Actual); Last update posted 2025-04-04 (Actual); Status verified 2024-09

CONDITIONS: Stroke; Aphasia
MeSH Terms: conditions — Stroke; Aphasia

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- active 1200-pulse cTBS group (Active Comparator): active 1200-pulse cTBS combined with speech language therapy
  Interventions: Device: active 1200-pulse continuous Theta Burst Stimulation
- active 2400-pulse cTBS group (Active Comparator): active 2400-pulse cTBS combined with speech language therapy
  Interventions: Device: active 2400-pulse continuous Theta Burst Stimulation
- active 3600-pulse cTBS group (Active Comparator): active 3600-pulse cTBS combined with speech language therapy
  Interventions: Device: active 3600-pulse continuous Theta Burst Stimulation
- sham 1200-pulse cTBS group (Sham Comparator): sham 1200-pulse cTBS combined with speech language therapy
  Interventions: Device: sham 1200-pulse continuous Theta Burst Stimulation
- sham 2400-pulse cTBS group (Sham Comparator): sham 2400-pulse cTBS combined with speech language therapy
  Interventions: Device: sham 2400-pulse continuous Theta Burst Stimulation
- sham 3600-pulse cTBS group (Sham Comparator): sham 3600-pulse cTBS combined with speech language therapy
  Interventions: Device: sham 3600-pulse continuous Theta Burst Stimulation

INTERVENTIONS:
Device: active 1200-pulse continuous Theta Burst Stimulation — Each patient will receive two 600-pulse cTBS stimulations per day, parted by a 15-minute rest period (a total of 1200 pulses daily), for 3-week treatment, with 5 consecutive workdays each week.
  Arms: active 1200-pulse cTBS group
Device: active 2400-pulse continuous Theta Burst Stimulation — Each patient will receive two 1200-pulse cTBS stimulations per day, parted by a 30-minute rest period (a total of 2400 pulses daily), for 3-week treatment, with 5 consecutive workdays each week.
  Arms: active 2400-pulse cTBS group
Device: active 3600-pulse continuous Theta Burst Stimulation — Each patient will receive two 1800-pulse cTBS stimulations per day, parted by a 50-minute rest period (a total of 3600 pulses daily), for 3-week treatment, with 5 consecutive workdays each week.
  Arms: active 3600-pulse cTBS group
Device: sham 1200-pulse continuous Theta Burst Stimulation — Each patient will receive two sham 600-pulse cTBS stimulations per day, parted by a 15-minute rest period (a total of 1200 pulses daily), for 3-week treatment, with 5 consecutive workdays each week.
  Arms: sham 1200-pulse cTBS group
Device: sham 2400-pulse continuous Theta Burst Stimulation — Each patient will receive two sham 1200-pulse cTBS stimulations per day, parted by a 30-minute rest period (a total of 2400 pulses daily), for 3-week treatment, with 5 consecutive workdays each week.
  Arms: sham 2400-pulse cTBS group
Device: sham 3600-pulse continuous Theta Burst Stimulation — Each patient will receive two sham 1800-pulse cTBS stimulations per day, parted by a 50-minute rest period (a total of 3600 pulses daily), for 3-week treatment, with 5 consecutive workdays each week.
  Arms: sham 3600-pulse cTBS group

SUMMARY:
The objective of this trial is to evaluate the effectiveness and safeness of different doses of continuous Theta Burst Stimulation (cTBS) over the right Superior Frontal Gyrus (SFG), guided by personalized Brain Function Sector (pBFS) technology, on language function recovery in patients with post-stroke aphasia.

DETAILED DESCRIPTION:
Increasing evidence suggests that rTMS has been effective in treating various psychological and neurological diseases, including treating post-stroke symptoms. Using the personalized brain functional sectors (pBFS) technique, investigators could precisely identify individualized brain functional networks and the personalized language-related stimulation site based on the resting-state functional MRI data. The current study proposes to conduct a double-blinded, randomized and parallel controlled design trial, to investigate the efficacy and safety of pBFS-guided personalized rTMS intervention in post-stroke aphasic patients.

Subjects will be randomly assigned to the following six groups: active 1200-pulse cTBS group, active 2400-pulse cTBS group, active 3600-pulse cTBS group, sham 1200-pulse cTBS group, sham 2400-pulse cTBS group, or sham 3600-pulse cTBS group. The allocation ratio will be 3:3:3:1:1:1. The stimulation protocol consisted of a 3-week treatment, with 5 consecutive workdays each week (totally 15 day-treatment). The stimulation procedure will be assisted with real-time neuronavigation to ensure its precision.

ELIGIBILITY:
Inclusion Criteria:

* The patient's age ranges from 35 to 75 years old (including 35 and 75 years old);
* Meet the diagnostic criteria for ischemic stroke (according to the guidelines developed by the American Heart Association/American Stroke Association in 2019 and the guidelines developed by the Neurology Branch of the Chinese Medical Association in 2018) or meet the diagnostic criteria for hemorrhagic stroke (according to the guidelines developed by the American Heart Association/American Stroke Association in 2022 and the guidelines developed by the Neurology Branch of the Chinese Medical Association in 2019) ，with lesions located in the left hemisphere, and a duration of illness ranging from 15 days to 6 months.
* Diagnosed as aphasia patient according to the Chinese version of Western Aphasia Battery (WAB), with a WAB-aphasia quotient of less than 93.8 points;
* First onset of stroke;
* Normal language function before the onset of stroke, and the patient's native language is Chinese with at least 6 years of education;
* Understand the trial and signed the informed consent form.

Exclusion Criteria:

* Combined dysarthria (NIHSS item 10 score ≥2 points);
* Aphasia caused by bilateral hemisphere stroke, brain tumor, traumatic brain injury, Parkinson's disease, motor neuron disease, or other diseases；
* Patients with implanted electronic devices such as cardiac pacemakers, cochlear implants, or other metal foreign bodies, or those with MRI contraindications such as claustrophobia or TMS treatment contraindications;
* History of epilepsy;
* Patient with concomitant severe systemic diseases affecting the heart, lungs, liver, kidneys, etc., and uncontrolled by conventional medication, as detected and confirmed through laboratory testing and examination;
* Patients with consciousness disorders (NIHSS 1(a) score ≥1);
* Patients with malignant hypertension;
* Patients with severe organic diseases, such as malignant tumors, with an expected survival time of less than 1 year;
* Patients with severe hearing, visual, cognitive impairment or inability to cooperate with the trial;
* Patients with severe depression, anxiety, or diagnosed with other mental illnesses that prevent them from completing the trial;
* Patients who have received other neuromodulation treatments such as TMS, transcranial electric stimulation, etc. in the 3 months prior to enrollment;
* Patients with a history of alcoholism, drug abuse, or other substance abuse;
* Patients with other abnormal findings that the researchers judge are not suitable for participation in this trial;
* Patients who are unable to complete follow-up due to geographical or other reasons;
* Women of childbearing age who are currently pregnant, breastfeeding, or planning or may become pregnant during the trial;
* Patients who are currently participating in other clinical trials.

Ages: 35 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2023-09-22 (Actual); Primary Completion 2025-09-22 (Estimated); Study Completion 2025-12-22 (Estimated)

PRIMARY OUTCOMES:
Change in the Western Aphasia Battery scores | baseline, end of the 3-week therapy
  The first four subsets of the WAB (Spontaneous Speech, Auditory verbal comprehension, Repetition, Naming and word finding) will be used to evaluate the participants' language ability impairments. A Chinese adapted version of WAB will be used. The scores from all four subsets will be calculated as an Aphasia Quotient (ranging from 0 to 100), with lower Aphasia Quotients indicating poorer language abilities.

SECONDARY OUTCOMES:
Change in the Western Aphasia Battery scores | baseline, end of the 5-day therapy, 90 days after treatment initiation
  The first four subsets of the WAB (Spontaneous Speech, Auditory verbal comprehension, Repetition, Naming and word finding) will be used to evaluate the participants' language ability impairments. A Chinese adapted version of WAB will be used. The scores from all four subsets will be calculated as an Aphasia Quotient (ranging from 0 to 100), with lower Aphasia Quotients indicating poorer language abilities.
Boston Diagnostic Aphasia Examination Severity Ratings | baseline，end of the 3-week therapy，90 days after treatment initiation
  The Boston Diagnostic Aphasia Examination (BDAE) Severity Ratings is a clinical tool used to evaluate the severity and type of aphasia in individuals. The assessment includes four domains: communication abilities, language content, speech sound production and response abilities.BDAE severity ratings range from level 0 to level 5, with lower scores indicating more severe aphasia.
Chinese-version Stroke and Aphasia Quality of Life Scale 39-generic version (SAQOL-39g) | baseline，end of the 3-week therapy，90 days after treatment initiation
  The SAQOL-39g is a quality of life assessment tool that is used to evaluate the impact of stroke and aphasia on a patient's quality of life. It consists of 39 items that cover a range of domains related to the patient's quality of life, such as communication, physical functioning, mood, and social support. The items are rated on a 5-point Likert scale ranging from "not at all" to "very much", with higher scores indicating better quality of life.

CONTACTS AND LOCATIONS:
Overall Officials: Hesheng Liu, PhD, Study Chair — Changping Laboratory
Locations (2):
- China (2):
  - Nanshi Hospital of Nanyang, Nanyang, Henan
  - The fifth Affiliated Hospital of Zhengzhou University, Zhengzhou, Henan